CLINICAL TRIAL: NCT01414816
Title: Betaferon® Regulatory Post-Marketing Surveillance
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14839; BF0814KR (Other: company internal)
Record Dates: First submitted 2011-07-13; First posted 2011-08-11 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Multiple Sclerosis; Clinically Isolated System
Keywords: Multiple Sclerosis; Clinical Isolated Syndrome (CIS)
MeSH Terms: conditions — Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — EOD, dosage frequency and duration will be decide by physicians.

SUMMARY:
To identify problems/questions about following items in the clinical practice using Betaferon

1. Unknown adverse event (especially serious adverse event)
2. Identification of adverse event occurred in the real practice
3. Factors that may affect the safety of drug
4. Factors that may affect the effectiveness of the drug

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of MS or CIS and decision taken by the physician to prescribe Betaferon
* Patients who have not participated in Betaferon regulatory Post Marketing Surveillance before.

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with local product information

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diagnosis of Multiple Sclerosis or Clinically Isolated Syndrome who have been or will be treated with Betaferon.
Sampling Method: Non-Probability Sample
Enrollment: 355 (Actual)
Dates: Start 2008-04; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Safety variables will be summarized using descriptive statistics based on adverse events. | Up to 6 months

SECONDARY OUTCOMES:
The efficacy data regarding prevention of relapse due to MS will be estimated based on the number of relapse. | During 6 month
Progression or aggravation to Multiple sclerosis (MS) will be identified based on the change of Expanded Disability Status Scale (EDSS) and the Magnetic Resonance Imaging (MRI) outcome. | 0, 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, South Korea